CLINICAL TRIAL: NCT06210373
Title: A Prospective, Multicentric, Randomized, Non-inferiority, Controlled, Open-label Clinical Investigation to Evaluate the Efficacy and Safety of the Use of Myrialen® Gel vs.Recugel®, Two Eye Gel Products Containing 5% Dexpanthenol, in Patients With Moderate to Severe Dry Eye Syndrome
Brief Title: Assessment of Efficacy and Safety of the Use of Two Eye Gel Products Containing 5% Dexpanthenol in Patients With Moderate to Severe Dry Eye Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS57-21-01
Record Dates: First submitted 2023-12-21; First posted 2024-01-18 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myrialen Gel Group (Experimental): Myrialen® gel: sterile ophthalmic gel containing 5% dexpanthenol
  Interventions: Device: Myrialen Gel
- Recugel Group (Active Comparator): Recugel®: sterile ophthalmic gel containing 5% dexpanthenol
  Interventions: Device: Recugel

INTERVENTIONS:
Device: Myrialen Gel — Myrialen Gel will be instilled as 1 drop per eye 3 times a day and one drop per eye before going to bed in the conjunctival sac for 30 days.In case of bilateral dry eye syndrome, both eyes will be treated. In case of monolateral dry eye syndrome, the decision to treat both eyes will be taken according to the Investigator's judgment.
  Other Names: Dexpanthenol 5%
  Arms: Myrialen Gel Group
Device: Recugel — Recugel will be instilled as 1 drop per eye 3 times a day and one drop per eye before going to bed in the conjunctival sac for 30 days.
  In case of bilateral dry eye syndrome, both eyes will be treated. In case of monolateral dry eye syndrome, the decision to treat both eyes will be taken according to the Investigator's judgment.
  Other Names: Dexpanthenol 5%
  Arms: Recugel Group

SUMMARY:
The prospective, multicentric, randomized, non-inferiority, controlled, open-label clinical investigation will evaluate the efficacy and safety of the use of Myrialen® gel vs.

Recugel®, two eye gel products containing 5% dexpanthenol, in patients with moderate to severe dry eye syndrome.

A total of 110 evaluable patients (55 in each treatment group), ≥18 years of age, will be required for data analysis. A total of 124 patients (62 in each treatment group) will be randomized to replace potential early withdrawals or non-evaluable patients.The primary objective of this investigation is to demonstrate non-inferior efficacy of Test Myrialen® gel over the Reference Recugel® in improving corneal and conjunctival surface state, assessed through slit lamp biomicroscopy examination, in patients with moderate to severe dry eye syndrome.

DETAILED DESCRIPTION:
There is scarce documentation in literature on the effects of dexpanthenol in the management of DED. In a randomized, double-blind, placebo-controlled study that evaluated the effect of dexpanthenol-containing artificial tears in 50 patients with dry eyes, patients receiving the active ingredient had significant improvement of disturbances of the corneal epithelial permeability (as measured by fluorophotometry and Schirmer test, Rose Bengal staining, TFBUT), compared to the dexpanthenol-free eyes drops. Despite the scarce literature documentation, the use of 5% dexpanthenol, which stimulates the processes of reparative regeneration and possesses an anti-inflammatory effect, is actually considered as one of the promising directions in the management of patients with DED. Dexpanthenol has also been developed as a component of a contact lens system that controls its release as osmoprotectant and moisturizing agent with the aim to reduce symptoms of ocular dryness.

Based on this background, this investigation has been designed to compare the effects of the investigational device Myrialen® gel with another device containing 5% dexpanthenol, i.e. Recugel® eye gel, in the treatment of patients with moderate to severe dry eye syndrome. In particular, the main objective of this investigation is to demonstrate that the test device Myrialen®gel will be non-inferior to the reference device Recugel® in improving corneal and conjunctival surface state.

ELIGIBILITY:
Inclusion Criteria:

1. Patient written informed consent to participate in the study obtained according to Good Clinical Practice (GCP);
2. Male and female patients aged ≥18 years;
3. Patients with new diagnosis of dry eye syndrome (according to Tear Film and Ocular Surface Society [TFOS] Dry Eye Workshop [DEWS] II definition), or previous diagnosis of dry eye syndrome not treated in the previous 15 days;
4. Diagnosis of dry eye syndrome performed through the following exams: slit lamp examination (SLE), Impact of Dry Eye on Everyday Living (IDEEL) questionnaire, tear (lacrimal) meniscus exam, Schirmer's test, Tear Film Break-Up Time (TFBUT), fluorescein and lissamine green staining of the cornea and conjunctiva (respectively). In case of bilateral dry eye syndrome, only the worst eye, defined as the eye with the higher severity of impairment according to theInvestigator's judgment based on the above exams, will be considered for assessments (although both eyes will be treated). In the case of bilateral dry eye syndrome with both eyes having the same level of impairment, the right eye will be considered for assessments by convention;
5. Sodium fluorescein and lissamine green staining score of the cornea and conjunctiva(respectively) ≥ 2 National Eye Institute (NEI) grid, defined as the sum of 5 areas per eye using a 0 (normal) to 3 (severe) scale) in the worst eye for the corneal staining and the sum of 6 areas per eye using a 0 (normal) to 3 (severe) scale in the worst eye for the conjunctival staining;
6. A Schirmer test value < 10 mm;
7. A TFBUT value ≥ 5 sec;
8. Patient able to comprehend the full nature and the purpose of the study, including possible risks and side effects, and subjects able to cooperate with the Investigator and to comply with the requirements of the entire study (including ability to attend all the planned study visits according to the time limits), based on Investigator's judgment;
9. Females of childbearing potential (i.e., not permanently sterilised - post hysterectomy or tubal ligation status - or not postmenopausal for at least one year) must have a negative urine pregnancy test result at Screening and must use an appropriate method of contraception for at least 30 days before inclusion in the study and during the whole study period, according to the definition in ICH M3 Guideline:

A highly effective method is defined as that which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Highly effective birth control methods include:

combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence.

Exclusion Criteria:

1. Any ocular disease other than dry eye syndrome requiring treatment with ophthalmological topical medications with re-epithelizing, trophic, anti-infective or anti-inflammatory effect (e.g. antibiotics, corticosteroids, gel re-epithelizing, platelet-rich plasma, autologous serum, medication with vitamin A, hyaluronic acid-based products) in either eye at the time of study enrolment and in the previous 30 days;
2. Any active ocular infection or active inflammation in either eye unrelated to dry eye syndrome;
3. Presence or history of any systemic or ocular disorder, condition or disease (with particular attention to malignancies and neuro-oncological diseases) that, according to Investigator's judgment, can interfere with the conduct of the required study procedures or the assessment of the efficacy or the interpretation of the study results or the incidence of adverse events;
4. Use of therapeutic or refractive contact lenses in either eye in the previous 20 days and at the time of study enrolment;
5. History of ocular surgery in either eye, excluding corneal refractive or cataract procedures, within 90 days of study enrolment;
6. Treatment with any other therapy that, according to Investigator's judgment, could interfere with the assessment of the efficacy or incidence of adverse events;
7. Hypersensitivity and/or allergy to any of Myrialen® gel and/or Recugel® ingredients;
8. Women pregnant or breastfeeding or women who could become pregnant and are not using effective contraception;
9. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the investigation;
10. Participation in another clinical investigation within the past 30 days or previous enrolment in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy assessment through National Eye Institute (NEI) total score compared to baseline | Day 30
  The NEI/Industry Workshop guidelines will be used as grading scale of the corneal and conjunctiva damage used. The cornea will be divided into five sectors (central, superior, inferior, nasal and temporal), each of which will be scored on a scale of 0-3, with a maximal score of 15. Both nasally and temporally, the conjunctiva will be divided into a superior paralimbal area, an inferior paralimbal area and a peripheral area with a grading scale of 0-3 and with a maximal score of 9 for the nasal and temporal conjunctiva.

SECONDARY OUTCOMES:
Efficacy assessment through National Eye Institute (NEI) total score compared to baseline | Day 7
  The NEI/Industry Workshop guidelines will be used as grading scale of the corneal and conjunctiva damage used. The cornea will be divided into five sectors (central, superior, inferior, nasal and temporal), each of which will be scored on a scale of 0-3, with a maximal score of 15. Both nasally and temporally, the conjunctiva will be divided into a superior paralimbal area, an inferior paralimbal area and a peripheral area with a grading scale of 0-3 and with a maximal score of 9 for the nasal and temporal conjunctiva.
Efficacy assessment through National Eye Institute (NEI) corneal score compared to baseline | Day 7 and Day 30
  The NEI/Industry Workshop guidelines will be used as grading scale of the corneal and conjunctiva damage used. The cornea will be divided into five sectors (central, superior, inferior, nasal and temporal), each of which will be scored on a scale of 0-3, with a maximal score of 15.
Efficacy assessment through National Eye Institute (NEI) conjunctival score compared to baseline | Day 7 and Day 30
  The NEI/Industry Workshop guidelines will be used as grading scale of the corneal and conjunctiva damage used. . Both nasally and temporally, the conjunctiva will be divided into a superior paralimbal area, an inferior paralimbal area and a peripheral area with a grading scale of 0-3 and with a maximal score of 9 for the nasal and temporal conjunctiva.
Assessment of Changes in impact of Dry Eye on Everyday living (IDEEL) questionnaire (symptom-bother and impact on daily life modules) from baseline | Day 30
  The IDEEL is divided into different sectionsa and only two will be considered in patient evaluation. The "Dry Eye Symptom-Bother" module includes 20 items: Item 1 from 0 "none of the time" to 4 "all of the time"; Items 2-from 1 "not at all" to 4 "very much". Score 0="I did not have this symptom / Not applicable"; and the "Dry Eye Impact on Daily Life" module composed of 3 sections: dry eye on daily living activities (9 items), emotional impact (12 items) and impact on work (6 items).Items 1-9 are scored on a 5-point Likert-like scale from 1 "all of the time" to 5 "none of the time". Items 10-21, 23-27 are scored on a 5-point Likert-like scale from 0 "all of the time" to 4 "none of the time". Item 22 is scored on a dichotomous scale: 1 "Yes", 0 "No". This item is not included in the calculation of the scores.
Assessment of Changes in Tear-Film Break-Up Time from baseline | Day 7 and Day 30
  The tear film is observed under cobalt-blue filtered light of the slit lamp biomicroscope and the time that elapses between the last blink and appearance of the first break in the tear film is recorded with a stopwatch (a break is seen as a dark spot in a sea of blue). TFBUT results of less than 10 seconds are consistent with dry eyes.
  The TFBUT will be measured twice during the first minute after the instillation of the fluorescein.
  If the 2 readings differ by more than 2 seconds a third reading will be taken. The TFBUT value will be the average of the 2 or 3 measurements.
Assessment of quantitative normalization of the tear film from baseline | Day 7 and Day 30
  Change in Schirmer's Test values from baseline. The Schirmer's test measures the quantity of total tear secretion, including reflex and basal tears, produced by the eye. A 35 mm x 5 mm size filter paper strip is used to measure the amount of tears that are produced over a period of 5 minutes. The wet portion of the strip is measured in millimeters. The test is done under ambient light. The patient is instructed to look forward and to blink normally during the course of the test. Normal mean test values range from 8 mm to 33 mm, but an accepted normal value is greater than 10 mm. Patients with dry eyes have wetting values of less than 5 mm in 5 minutes.
Assessment of qualitative normalization of the tear film from baseline | Day 30
  Changes will be evaluated through the tear meniscus height. The tear (lacrimal) meniscus examination is conducted using slit-lamp biomicroscopy (narrow slit and low intensity light) and observing the tear (lacrimal) meniscus height. Values are considered normal if within the 0.3 to 0.5-mm range.
Assessment of changes in visual acuity from baseline | Day 30
  Visual function will be assessed by distance visual acuity measurement. Both uncorrected distance visual acuity (UNVA, vision with no extraocular optical correction) and best corrected distance visual acuity (BCVA, defined as obtained with the best possible refractive correction) will be measured using the Snellen chart. Visual acuity values will be expressed in decimal, fraction or logMAR. All assessments will be performed using standard charts and procedures at specified visual angle, illumination and contrast. Current refraction will be determined prior to visual acuity testing to obtain best-corrected vision
Assessment of incidence of treatment-emergent adverse events | Day 30
  Safety and tolerabiltiy will be assessed through the analysis of Incidence and nature of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs); Incidence and nature of Adverse Device Effects (ADEs) and serious ADEs (SADEs) during the entire investigation duration; Incidence and nature of Investigational Medical Device Deficiencies (IMDDs) during the entire investigation duration.

OTHER OUTCOMES:
Changes in confocal microscopy of density of dendritic cells from baseline | Day 30
  The changes will be evaluated through the use of confocal microscopy. The density of dendritic cells at the level of the sub-epithelial basal membrane evaluated in the central cornea (number of cells/mm2) will be evaluated according to single-layer epithelium, two cellular layers evidenced, more than two cellular layers evidenced.
Changes in confocal microscopy in stratification of the epithelium from baseline | Day 30
  The changes will be evaluated through the use of confocal microscopy. The stratification of the epithelium will be evaluated according to single-layer epithelium, two cellular layers evidenced, more than two cellular layers evidenced.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Mastropasqua, MD, Principal Investigator — Ospedale SS. Annunziata- Università degli studi G. d'Annunzio-Chieti
Locations (3):
- Italy (3):
  - Ospdale SS.Annunziata-Università degli Studi G.d'Annunzio, Chieti, Pescara
  - Università degli studi Federico II, Napoli
  - Humanitas Gradenigo, Torino

IPD SHARING:
Plan to Share IPD: No